CLINICAL TRIAL: NCT02506387
Title: Belgian Mitraclip Registry
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, M Claeys, Prof dr, Universiteit Antwerpen
Other Study IDs: BEL 0
Record Dates: First submitted 2015-07-19; First posted 2015-07-23 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mitraclip patients: Patients with severe mitral regurgitation in whom decision for mitraclip implantation was made by the heart team.
  Interventions: Device: mitraclip

INTERVENTIONS:
Device: mitraclip — The decision to implant mitraclip is not part of this observational study but is made by the heart-team.

SUMMARY:
The primary objective of the registry is to investigate and follow all patients treated with the MitraClip System in Belgium. This information is intended to contribute to decision making with regards to MitraClip therapy selection in patients with mitral regurgitation: (a) by establishing the clinical value of the MitraClip therapy in the continuum of care; and (b) by providing practical information that will allow physicians to make therapeutic decisions, assist hospitals to make purchasing decisions, and assist insurers/government in making coverage decisions.

In addition national data will be shared with European registries in order to increase the knowledge about the efficacy of this new technique.

ELIGIBILITY:
Inclusion Criteria:

* severe mitral regurgitation
* symptomatic (NYHA class>1) despite optimal medical therapy
* suitable anatomy for mitraclip implantation
* too high risk for cardiac surgery

Exclusion Criteria:

* <1 year life expectancy

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with symptomatic severe mitral regurgitation at too high risk voor cardiac surgery and with suitable anatomy for mitraclip implantation
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2015-01; Primary Completion 2023-01 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
residual mitral regurgitation (MR) post mitraclip | at day 3-5 post mitraclip implantation
  MR grade 1 tot 4, as assessed on echocardiography
cardiac mortality | 2 years
surgical mitral valve intervention | 2 years
hospitalization for heart failure | 2 years
  heart failure as primary reason of hospitalization

SECONDARY OUTCOMES:
pericardial effusion | day 1-2 after mitraclip implantation
  peri-procedural pericardial effusion with hemodynamic impact as assessed on echocardiography
change in New York Heart Association (NYHA) classification | 2 years
  NYHA 1-4 as assessed by the clinician at baseline and 1 month, 6 month, 1 year and 2 year after mitraclip implantation
distance during 6 min walking test | 1 year
  distance expressed in meters assessed baseline, 6 month and 1 y after mitraclip implantation.
Left ventricular (LV) remodeling | 6 month
  echocardiac evaluation of LV end diastolic volume (LVEDV) with calculation of LV remodeling according to following formula: (LVEDV at six month - LVEDV baseline)/ LVEDV baseline
Acute renal failure requiring dialysis | up to one month after mitraclip implantation
  Acute renal failure requiring dialysis
urgent surgical mitral valve intervention | within 24h after procedure
  urgent surgical mitral valve intervention
Change in Left ventricular ejection fraction (LVEF) | 6 month
  echocardiac evaluation of LV end systolic volume ( LVESV) and LV end diastolic volume (LVEDV) with calculation of LVEF according to following formula: (LVEDV - LVESV)/ LVEDV . LVEF measured at baseline and 6 month after mitraclip implantation

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University hospital Antwerp, Edegem, Antwerp
  - OLV Aalst, Aalst